CLINICAL TRIAL: NCT03275636
Title: A Randomized Controlled Trial Comparing Outcome After Hematopoietic Cell Transplantation From a Partially Matched Unrelated Versus Haploidentical Donor
Brief Title: Haploidentical Donor vs mMUD in Hematological Malignancies
Acronym: HAMLET
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: DKMS gemeinnützige GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DKMS-16-01; 2015-005399-12 (EudraCT Number)
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: AML; ALL; MDS
Keywords: Haploidentical; mismatched unrelated donor; hematopoietic stem cell transplantation; donor comparison

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haploidentical donor (Experimental): Peripheral blood stem cells from Haploidentical donor
  Interventions: Biological: Peripheral blood stem cells
- partially matched unrelated donor (Active Comparator): Peripheral blood stem cells from unrelated donor with a single allele or antigen mismatch at HLA-A, -B, -C, or -DRB1 and no concurrent DQB1 mismatch (9/10) shown by confirmatory typing
  Interventions: Biological: Peripheral blood stem cells

INTERVENTIONS:
Biological: Peripheral blood stem cells — Hematopoietic stem cell transplantation with PBSC
  Other Names: PBSC

SUMMARY:
The goal of this trial is to compare the outcome after partially matched (single mismatch) unrelated donor transplantation with haploidentical transplantation in a randomized controlled setting.

DETAILED DESCRIPTION:
For patients with an indication for allogeneic HCT, the search for a stem cell donor is a challenge. 20% of patients who need an allograft have an HLA-identical sibling available, and for approximately 70% of the remaining patients, a suitable, HLA-well-matched (10/10), unrelated volunteer can be found. For the remaining patients, partially matched (single mismatch) unrelated donors or haploidentical donors are alternative options.

Recently published retrospective single center and registry studies suggest comparable outcomes for HCT from unrelated donors matched at HLA -A, -B, -C, and -DRB1 and haploidentical donors. The number of haploidentical HCT evaluated in these studies was still relatively small and a selection bias for the retrospective comparisons cannot be excluded.

The goal of this trial is to evaluate overall survival of patients with high-risk AML, ALL or MDS after partially matched unrelated or haploidentical donor transplantation..

ELIGIBILITY:
Inclusion criteria

1. Eligible diagnoses are listed below:

   AML with adverse risk genetic abnormalities (according to the ELN guidelines)1. AML with intermediate genetic abnormalities (according to ELN guidelines) either in first complete remission, after relapse, or by chemotherapy-refractory disease.

   AML with favourable genetic abnormalities (according to ELN guidelines) after relapse or by chemotherapy-refractory disease, except APL.

   AML with undefined genetic risk classification after relapse or with chemotherapy-refractory disease.

   AML arising from myelodysplastic syndrome (MDS) or a myeloproliferative neoplasia, except if favourable genetic abnormalities (according to ELN guidelines) are present.

   Therapy-related myeloid neoplasia except if favorable genetic abnormalities (according to ELN guidelines) are present.

   MDS with high risk or very high risk disease (according to the IPSS-R score)2.

   First CR of high-risk ALL, defined by one or more of these:
   * Early or mature T-ALL (CD1a negative).
   * Pro B-ALL with t(4v;11); KMT2A-rearrangements.
   * Presence of BCR-ABL and/or t(9;22).
   * Persistence of minimal residual disease after the second induction course. ALL with or without complete remission after salvage therapy following poor response to induction therapy.

   ALL after haematological or molecular relapse.
2. Fit for transplant according to physician judgement.
3. No history of cardiac disease and absence of active symptoms, otherwise, documented left ventricular ejection fraction ≥40%.
4. No history of chronic pulmonary disease and absence of dyspnea. Otherwise, documented diffusion lung capacity for carbon monoxide (DLCO) ≥40% or FEV1/FVC ≥ 50% despite appropriate treatment
5. Availability of ≥1 unrelated donor with a single allele or antigen mismatch at HLA-A, -B, -C, or -DRB1 and no concurrent DQB1 mismatch (9/10) shown by confirmatory typing.
6. Availability of at least one haploidentical donor meeting the following criteria:

Donor is a biologic parent / child of the patient, or haploidentity has been confirmed for patient's relatives by HLA-Typing.

The donor has expressed his/her will to donate and has no contraindications against a stem cell donation by medical history.

Donor age is ≥18 years and ≤75 years.

Exclusion criteria

1. Relapse or graft failure after a first allogeneic transplantation.
2. Thymic ALL in first complete remission.
3. Severe organ dysfunction defined by either of the following three criteria:

   Patients who receive supplementary continuous oxygen. Serum bilirubin >1.5 x ULN (if not considered Gilbert-Syndrome) or ASAT/ALAT >5 x ULN.

   Estimated Glomerular Filtration Rate (GFR) < 40 mL/min
4. Uncontrolled infection at the time of enrollment.
5. Pregnant or breast-feeding women.
6. An HLA-identical sibling donor or 8/8 (HLA-A, -B, -C, or -DRB1) matched unrelated donor is available and suitable to donate prior to randomization.
7. Men unable or unwilling to use adequate contraception methods from enrollment to minimum of six months after the last dose of chemotherapy.
8. Women of childbearing potential except those who fulfill the following criteria: Post-menopausal or post-operative or continuous and correct application of a contraception method with a Pearl Index <1% or sexual abstinence or vasectomy of the sexual partner.
9. Simultaneous participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival calculated from the time of randomization will be the primary endpoint of this trial. Death from any reason will be considered as event.

SECONDARY OUTCOMES:
Engraftment rate | day 56
  Engraftment
Immune-reconstitution rate | day56
  Immune-reconstitution rate
Infections | 2 months after HCT
  Severe infections rate
Event Free Survival | 1 year
  Event Free Survival
Graft vs Host Disease | 1 year
  Graft vs Host Disease rate
Graft vs Host Disease-free survival | 1 year
  Graft vs Host Disease-free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, Prof Dr med, Study Chair — Universtitätsklinikum Dresden
Locations (9):
- Germany (9):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen